CLINICAL TRIAL: NCT03971682
Title: The Efficacy of a Compassion Focused Therapy-based Intervention in Detained Youth: A Clinical Trial
Brief Title: The Efficacy of a Compassion Focused Therapy-based Intervention in Detained Youth
Acronym: PSYCOMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Diana Ribeiro da Silva, Principal investigator, University of Coimbra
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CINEICC-1-DRS; SFRH/BD/99795/2014 (Other Grant/Funding Number: Portuguese Foundation for Science and Technology (FCT)); POCI-01-0145-FEDER-016724 (Other Grant/Funding Number: FEDER, COMPETE 2020, FCT)
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Psychopathic Personality Trait; Conduct Disorder; Delinquency
Keywords: Conduct Disorder; Compassion Focused Therapy; Detained Youth; Psychopathic Traits; PSYCHOPATHY.COMP
MeSH Terms: conditions — Conduct Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental - PSYCHOPATHY.COMP program. (Experimental): The PSYCHOPATHY.COMP is a structured individual program for detained youth. This program is based on Compassion Focused Therapy (CFT), which conceptualizes antisocial behavior and psychopathic traits as evolutionary rooted responses to deal with harsh rearing scenarios. The ultimate goal of the PSYCHOPATHY.COMP is to develop a compassionate motivation in these youth.
  PSYCHOPATHY.COMP consists of 20 individual sessions, each lasting about 60 minutes, which run on a weekly basis. Sessions must be carried out by therapists skillful in CFT. Sessions are grouped into four modules: (1) The basics of our mind; (2) Our mind according to CFT; (3) Compassionate Mind Training; and (4) Recovery, relapse prevention, and finalization.
  The treatment group attended the PSYCHOPATHY.COMP program in addition to the Treatment As Usual (TAU) delivered at Portuguese juvenile detention facilities.
  Interventions: Behavioral: PSYCHOPATHY.COMP program.; Other: Treatment As Usual - TAU
- Treatment As Usual - TAU (Active Comparator): Treatment As Usual:
  Subjects in this group received Treatment As Usual in Portuguese juvenile detention facilities (school frequency, token economy system for behavior control, frequency of a structured cognitive-behavioral group program, as well as individualized counseling sessions delivered by psychologists from the juvenile justice system) and did not attend the PSYCHOPATHY.COMP program.
  Interventions: Other: Treatment As Usual - TAU

INTERVENTIONS:
Behavioral: PSYCHOPATHY.COMP program. — The PSYCHOPATHY.COMP program is a structured individualized program for detained youth based on Compassion Focused Therapy, aimed to develop a compassionate motivation in these youth.
  Treatment As Usual Treatment As Usual (TAU) in Portuguese juvenile detention facilities is primarily aimed to increase educational and professional qualifications, as well as to promote behavioral regulation.
  Arms: Experimental - PSYCHOPATHY.COMP program.
Other: Treatment As Usual - TAU — Treatment As Usual (TAU) in Portuguese juvenile detention facilities is primarily aimed to increase educational and professional qualifications, as well as to promote behavioral regulation.

SUMMARY:
This non-randomized controlled trial with a control group aimed to assess the efficacy of a 20-session individualized Compassion Focused Therapy-based intervention, the PSYCHOPATHY.COMP, in reducing psychopathic traits (primary outcomes), aggression, shame, emotion regulation problems, and fears of compassion, as well as in increasing social safeness, self-compassion, and compassion towards others (secondary outcomes). The PSYCHOPATHY.COMP's impact on psychophysiological (i.e., Heart Rate/Heart Rate Variability) and behavioral indicators (i.e., number disciplinary infractions and number of days in punishment) were also tested, in order to ascertain if changes observed in self-report questionnaires were reflected in more adjusted psychophysiological and behavioral patterns. Mental Health disorders, as well as the number of Conduct Disorder criteria, were also tested as moderators of treatment effects.

DETAILED DESCRIPTION:
This was a non-randomized controlled trial with a control group carried out in the six Portuguese juvenile detention facilities aimed to test the efficacy of an individual Compassion Focused-based intervention (the PSYCHOPATHY.COMP program) in detained youth.

The ethics committee of the Faculty of Psychology and Educational Sciences of the University of Coimbra, the National Data Protection Agency, and the Portuguese Ministry of Justice approved the study's procedures. Portuguese juvenile detention facilities usually have no more than 150 detained youth (about 30 youth per juvenile detention facility), facing 6 to 36 months of detention, around 10 youth enter and leave Portuguese juvenile detention facilities per month, which makes it difficult to randomly assign participants to conditions. To try to minimize this roadblock and to maximize time and human resources, the research team opted to assign the first 60 youth entering in the juvenile detention facilities during the research period to the treatment group and the following 60 youth to the control group. Participants in the treatment group attended the PSYCHOPATHY.COMP program for about 6 months in addition to the treatment as usual (TAU) delivered at Portuguese juvenile detention facilities. The TAU in Portuguese juvenile detention facilities is primarily aimed to increase educational and professional qualifications, as well as to promote behavioral regulation and encompasses: school frequency, a token economy system for behavior control, the frequency of a cognitive-behavioral group program (the GPS-Growing Pro-Social; Rijo et al., 2007) and individual counseling sessions delivered by psychologists from the juvenile justice system (the treatment group would not attend these sessions). Participants in the control group received TAU, including the individual counseling sessions delivered by psychologists from the juvenile justice system, and did not attend the PSYCHOPATHY.COMP during the research period.

Researchers invited detained youth to voluntarily participate in the study, explained its goals, and presented a brief overview of the intervention program. Confidentiality and anonymity were guaranteed. It was also explained to detained youth that their participation in the study would not impact on their sentencing/school grades in any possible way. Participants who agreed to participate gave written informed consent, in addition to their parents/legal guardians' written consent, and completed the baseline assessment. Participants in the control group were informed that they would benefit from the individualized counseling sessions by the psychologists from the juvenile detention facilities.

Participants in the treatment group were assessed before the first session of the program (baseline assessment), right after its terminus (i.e., post-treatment assessment - about 6 months after the baseline assessment), and 6 months after PSYCHOPATHY.COMP completion (follow-up assessment). Participants in the control group were assessed with the same time intervals. Independent research assistants blind to condition assignment participated in data collection. Respondent-specific codes were used to link the data from one time-point to the next one. These researchers received intensive training on the assessment measures and had supervision sessions with a senior researcher during data collection.

PSYCHOPATHY.COMP's therapists were three psychologists, who had at least six years of clinical experience as well as intensive training and experience in delivering the PSYCHOPATHY.COMP program to young offenders. Moreover, therapists received weekly supervision by a senior CFT expert during the time PSYCHOPATHY.COMP was run in juvenile detention facilities. Therapist and youth rated every session and 5% of the sessions were observed by independent raters in order to assess treatment integrity. Finally, the program's structured and manualized design also accounted for integrity, at least partially.

ELIGIBILITY:
Inclusion Criteria:

* Detained youth aged between 14 and 18 years old
* Presence of Conduct Disorder as the main diagnosis (MINI-KID)

Exclusion Criteria:

* Non-Portuguese speaking (to avoid communication issues);
* Remaining in the juvenile detention facility less than 12 months since the beginning of the program (taking into account PSYCHOPATHY.COMP length and assessment period)
* Presence of cognitive disabilities (because PSYCHOPATHY.COMP is not suitable for cognitively-impaired youth)
* Presence of psychotic symptoms (the experiential exercises used in the program are contraindicated for psychotic patients)
* Presence of autism spectrum disorders (because PSYCHOPATHY.COMP was not designed considering the social impairments of these youth).

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change of psychopathic traits | baseline; 6 months, 12 months
  Participants reported on the Youth Psychopathic Traits Inventory-Short (YPI-S; Van Baardewijk et al. 2010). The YPI-S is an 18-item self-report questionnaire, which assesses psychopathic traits in youth via ratings within three different factors: Grandiose-Manipulative (GM); Callous-Unemotional (CU), and Impulsive-Irresponsible (II). Each factor is estimated by a set of six items; each item is rated on a four-point scale (1 = "Does not apply at all" to 4 = "Applies very well").This assessment was carried out by researchers, who received training in this self-report measures.
Change psychopathic traits | baseline; 6 months, 12 months
  Participants reported on the Proposed Specifiers for Conduct Disorder (PSCD; Salekin & Hare, 2016). The PSCD is a 24-item self-report questionnaire, which assesses the above mentioned psychopathic traits, as well as antisocial behavior. Each factor is estimated by a set of six items; each item is rated on a three-point scale (0 = "False" to 2 = "True"). This assessment was carried out by researchers, who received training in this self-report measures.

SECONDARY OUTCOMES:
External Shame | baseline; 6 months, 12 months
  Participants reported on a questionnaire of external shame, the Other as Shamer Scale Brief-Adolescent version (OASB-A; Vagos et al., 2016b). The OASB-A is an 8-item self-report scale that measures external shame, i.e., a subject's perception of being negatively judged by others. Items are rated on a five-point frequency scale (0= "Never"; 4-"Almost Always"), reporting how frequently one experiences the feelings described in each statement. This assessment was carried out by researchers, who received training in the self-report measure.
Social Safeness and Pleasure | baseline; 6 months, 12 months
  Participants reported on a questionnaire of social safeness and pleasure, the Social Safeness and Pleasure Scale (SSPS; Cook, 1996). The SSPS is an 11-item self-report scale that measures social safeness, i.e., the extent to which individuals feel a sense of acceptance and connectedness in their social relationships. Items are rated on a 5-point scale (1 = "Almost never" to 5 = "Almost all the time"). This assessment was carried out by researchers, who received training in the self-report measure.
Self-Compassion | baseline; 6 months, 12 months
  Participants reported on a questionnaire of self-compassion, the Self-Compassion Scale (SCS; Neff 2003a). The SCS is a 26-item self-report scale, which assesses trait levels of self-compassion. It includes items that measure how often people respond to feelings of inadequacy or suffering with self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. Responses are given on a 5-point scale from (1 = "Almost Never" to 5 = "Almost Always"). This assessment was carried out by researchers, who received training in the self-report measure.
Compassion | baseline; 6 months, 12 months
  Participants reported on a questionnaire of compassion, the Compassion Scale (CS; Pommier, 2011). The CS is a 24-item self-report questionnaire that measures compassion for others, and it is composed by six subscales: Kindness; Common Humanity; Mindfulness; Indifference; Separation, and Disengagement. Participants rate each item according to how frequently they feel and act towards others, using a five-point scale (1 = "Almost Never" to 5 = "Almost Always"). This assessment was carried out by researchers, who received training in the self-report measure.
Fears of Compassion | baseline; 6 months, 12 months
  Participants reported on a questionnaire of fears of compassion, the Fears of Compassion Scale (FCS; Gilbert, McEwan, Matos, & Rivis, 2011). The FCS is a three-section measure that assesses fears related to giving and receiving compassion and fears of self-compassion. Items are rated on a 5-point scale (0 = "Totally disagree" to 4 = "Totally Agree"). This assessment was carried out by researchers, who received training in the self-report measure.
Emotion Regulation | baseline; 6 months, 12 months
  Participants reported on a questionnaire of emotion regulation, the Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004). The DERS is a 36-item self-report measure that assesses individuals' typical levels of emotion dysregulation across six separate domains: non-acceptance of negative emotions, inability to engage in goal-directed behaviors when experiencing negative emotions, difficulties controlling impulsive behaviors when experiencing negative emotions, limited access to emotion regulation strategies perceived as effective, lack of emotional awareness, and lack of emotional clarity. Items are scored on a 5-point scale (1 = "Almost never" to 5 = "Almost Always"). This assessment was carried out by researchers, who received training in the self-report measure.
Heart Rate/Heart Rate Variability | baseline; 6 months, 12 months
  Psychophysiological measures of HR/HRV of the participants were collected throughout an experimental procedure designed in accordance to the conceptual model of Compassion Focused Therapy. This assessment was carried out by researchers, who received specific training.
Disruptive Behavior | from baseline to 6 months' follow-up
  To assess behavior regulation during the research period, a grid was developed to collect the following data from participants' record files: number of disciplinary infractions and number of days in punishment.

OTHER OUTCOMES:
Psychopathology | Baseline
  Participants were interviewed with the Mini-International Neuropsychiatric Interview for Children and Adolescents (MINI-KID; Sheehan et al., 2010). The MINI-KID is a structured clinical diagnostic interview, which assesses DSM disorders in children and adolescents. This assessment was carried out by researchers who had special training in the diagnosis of psychopathological disorders and previous experience administering the MINI-KID interview.
Recidivism Risk Assessment | Baseline
  Recidivism risk was assessed through the Youth Level of Service/Case Management Inventory (YLS/CMI; Hoge, Andrews, & Leschied, 2002). This assessment was completed by a probation officer. The YLS/CMI is a 42-item checklist, which assesses eight different risk factors/needs: Prior and Current Offenses/Disposition, Family Circumstances/Parenting, Education/Employment, Peer Relations, Substance Abuse, Leisure/Recreation, Personality/Behavior, and Attitudes/Orientation. Each item is scored dichotomously (present/absent). Each response in the affirmative receives a point towards the respective factor score and also to the total score (i.e., the sum of all eight risk/need scores). In this trial, the total risk score of the YLS/CMI was used as a measure of recidivism risk. Based on the total score, youth can be categorized into four levels of recidivism risk: low (0-8 points), moderate (9-22 points), high (23-34 points), or very high (35-42 points).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rijo, PhD, Principal Investigator — CINEICC
Locations (1):
- Faculty of Psychology and Educational Sciencies, University of Coimbra, Coimbra, Portugal

REFERENCES:
- [Derived] Sousa R, Ribeiro da Silva D, Petrocchi N, Gilbert P, Rijo D. At the heart of change: Differences in young offenders' HRV patterns after the delivery of the PSYCHOPATHY.COMP program. Front Psychiatry. 2023 Jan 10;13:1032011. doi: 10.3389/fpsyt.2022.1032011. eCollection 2022. PMID 36704737
- [Derived] Rijo D, Ribeiro da Silva D, Brazao N, Paulo M, Ramos Miguel R, Castilho P, Vagos P, Gilbert P. Promoting a compassionate motivation in detained youth: A secondary analysis of a controlled trial with the PSYCHOPATHY.COMP program. Personal Disord. 2023 Mar;14(2):223-236. doi: 10.1037/per0000594. Epub 2022 Jul 28. PMID 35901377
- [Derived] Ribeiro da Silva D, Rijo D, Brazao N, Paulo M, Miguel R, Castilho P, Vagos P, Gilbert P, Salekin RT. The efficacy of the PSYCHOPATHY.COMP program in reducing psychopathic traits: A controlled trial with male detained youth. J Consult Clin Psychol. 2021 Jun;89(6):499-513. doi: 10.1037/ccp0000659. PMID 34264698